CLINICAL TRIAL: NCT04527848
Title: Comparison of Two Intraocular Gas Injection Techniques in Macula Hole Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Rodrigo Pessoa Cavalcanti Lira, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12347319.9.0000.8807
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Macular Holes
Keywords: macular holes; Injections, Intra-Ocular; gases
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The individuals were randomized in a 1: 1: 1: 1 ratio. Block sizes of 4 individuals stratified according to gas type were used (SF6 or C3F8). In each block, two individuals were allocated to each group (0.9-1.0 mL of 100% gas or 15-20 mL of 20% gas).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- small amount of undiluted C3F8 (Experimental)
  Interventions: Drug: small amount of undiluted C3F8
- large amount of diluted C3f8 (Active Comparator)
  Interventions: Drug: small amount of undiluted C3F8
- small amount of undiluted SF6 (Active Comparator)
  Interventions: Drug: small amount of undiluted C3F8
- large amount of diluted SF6 (Active Comparator)
  Interventions: Drug: small amount of undiluted C3F8

INTERVENTIONS:
Drug: small amount of undiluted C3F8 — vitrectomy followed by peeling of the internal limiting membrane and, after that, intraocular gas injection

SUMMARY:
To undertake a prospective randomized clinical trial of vitrectomy and gas tamponade to treat macular hole, utilizing a small amount of undiluted C3F8 (perfluoropropane) versus a large amount of diluted C3F8 versus a small amount of undiluted SF6 (sulfur hexafluoride) versus a large amount of diluted SF6.

ELIGIBILITY:
Inclusion Criteria:

* pseudophakia
* without previous vitreoretinal surgery
* diagnosed with a full-thickness macula hole on the optical coherence tomography exam.
* duration of symptoms less than 6 months
* inform consent

Exclusion Criteria:

* ocular trauma
* allergy to any of the products used in the study,
* need to travel by plane in the first 60 postoperative days
* myopia over 6 diopters or axial diameter over 26 mm
* retinal dystrophies
* retinal detachment
* abnormal eye shape
* glaucoma
* diabetic retinopathy or other eye comorbidities.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Gas duration | up to 60 days
  duration of intraocular gas
macula hole closure | 26 weeks
  closure of the macular hole after the primary surgical procedure

SECONDARY OUTCOMES:
visual acuity | preoperative, 26 weeks
  corrected distance visual acuity
intraocular pressure | preoperative, 1 day, 26 weeks
  intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo PC Lira, PhD, Principal Investigator — UFPE
Locations (1):
- UFPE Ophthalmology, Recife, Pernambuco, Brazil